CLINICAL TRIAL: NCT04915417
Title: A Pilot Study to Assess the Safety and Feasibility of Neoadjuvant Stereotactic Ablative Radiotherapy for Pancreatic Ductal Adenocarcinoma
Brief Title: Neoadjuvant Stereotactic Ablative Radiotherapy for Pancreatic Ductal Adenocarcinoma
Acronym: ANSR-PDAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 118543
Record Dates: First submitted 2021-05-14; First posted 2021-06-07 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Resectable Pancreatic Adenocarcinoma; Borderline Resectable Pancreatic Adenocarcinoma
Keywords: Stereotactic Ablative Body Radiation Therapy; Neoadjuvant; Pancreatic Adenocarcinoma; Hybrid PET/MRI; CT Perfusion; Blood Proteomics; Immunomodulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resectable Pancreatic Ductal Adenocarcinoma (PDAC) (Experimental): 10 Resectable PDAC patients will receive a hybrid PET/MRI before SABR and DCE-CT before SABR, 6 hours after the first SABR fraction, and 4 weeks after the last fraction of SABR (before surgery)
  Interventions: Radiation: Stereotactic Ablative Body Radiotherapy (SABR)
- Borderline Resectable Pancreatic Ductal Adenocarcinoma (PDAC) (Experimental): 20 Borderline Resectable PDAC patients will receive a DCE-CT scan prior to neoadjuvant chemotherapy, a PET/MRI and DCE-CT after neoadjuvant chemotherapy and before SABR, DCE-CT at 6 hours after the first SABR fraction, and 4 weeks after the last fraction of SABR (before surgery)
  Interventions: Radiation: Stereotactic Ablative Body Radiotherapy (SABR)

INTERVENTIONS:
Radiation: Stereotactic Ablative Body Radiotherapy (SABR) — Patients will receive 27-30 Gy in 3 fractions to the planning target volume (PTV) with a simultaneous in-field boost to the metabolically active areas of the gross tumor volume (GTV) to a maximum of 45 Gy. Patients will be treated every other day.

SUMMARY:
Pancreatic cancer (PC) is expected to be the third leading cause of cancer death in Canada in 2019 [1]. Localized pancreatic cancer may be classified as resectable, borderline resectable, or locally advanced. To date, radical surgical resection and adjuvant treatment provide the greatest chance of long-term disease control and overall survival [2,3]. Despite this favourable group, the five-year survival rates are approximately 20% [4].

Neoadjuvant therapy (NAT) for resectable pancreatic cancer (RPC) has been widely accepted for the management of borderline resectable PC (BRPC) to increase the likelihood of achieving R0 resection [4-7]. However, to date, NAT for RPC is still an area of debate due to the lack of large prospective randomized controlled trials that compare this technique to surgery plus adjuvant therapy.

Stereotactic ablative radiation therapy (SABR) uses modern radiotherapy planning and targeting technologies to precisely deliver larger, ablative doses of radiotherapy in 1-8 fractions. The role of SABR in RPC has yet to be fully established. The typical goal of radiation therapy in the neoadjuvant setting is to improve local control and increase R0 resection rates. However, there are still concerns about the timing of surgery after SABR and any implementation should be evaluated for safety.

Treatments inherently changes the tumour and can cause immunomodulatory effects. SABR has anti-neoplastic effects both directly on the tumour and by its interactions with the immune system. In addition to the direct DNA damage, it is felt that SABR also increases T-cell priming, antigen production and presentation. Pancreatic cancer's dense, collagen rich stroma has prevented patients from receiving the same benefits of checkpoint inhibition that have been achieved in other cancer sites.

DETAILED DESCRIPTION:
Goals: The primary goals of this study are to evaluate the safety and feasibility of neoadjuvant SABR patients with surgical PC. This proposal is specifically intended to strengthen the correlative sciences evaluating pre- and post-treatment tissue samples and serial plasma samples evaluating the immunomodulatory effects of neoadjuvant SABR.

Population: Patients with upfront resectable pancreatic adenocarcinoma (RPC) with a plan to proceed directly to curative surgery or borderline resectable pancreatic adenocarcinoma (BRPC) with a plan for neoadjuvant FOLFIRINOX chemotherapy with the hopes of then proceeding to a curative surgical resection will be accrued.

Objectives and Endpoints: The primary objective is to determine the safety and feasibility of neoadjuvant SABR in patients with PC. Secondary objectives include (1) determining the tumor perfusion with serial dynamic contrast enhanced CT imaging studies; (2) evaluating serial peripheral blood samples for changes in markers of inflammation or immune activation using O-link's plasma-based proteomics platform; (3) T-cell receptor (TCR) sequencing from RNA isolated from the buffy coat from serial whole blood samples; (4) Digital spatial profiling on FFPE samples from pre-treatment biopsy tissue and post-treatment surgical resection samples to examine CD3, CD8, PD-L1 expression and other markers of immunomodulation; (5) RNA sequencing (RNA-Seq) will be conducted on pre- and post-treatment samples to examine the gene expression profile within specific areas of the tumor environment; (6) examining the influence of SABR on classic biomarkers such as CEA and CA19-9.

Methodology: Upfront RPC (n=10) and BRPC (n=20) with the expectation of approximately 10 participants receiving neoadjuvant SABR on study.

Imaging Studies: Patients in both arms will receive both a hybrid PET/MRI scan and a dynamic contrast enhanced (DCE-CT) scan prior to SABR to define high metabolic regions (using 18F-FDG PET), define the whole tumour border (using MRI), and to define baseline perfusion parameters such as blood flow, blood volume, permeability surface, and mean transit time (using DCE-CT). This information will be used to define regions that will receive high doses of radiation therapy. These patients will also receive a DCE-CT scan six hours after the first of three radiation treatments and 4 weeks following SABR (before surgery) to investigate changes in blood flow.

ELIGIBILITY:
Inclusion Criteria (Both Arms):

* Age 18 or older
* Able to provide informed consent
* Histologically confirmed primary pancreatic cancer, or willing to undergo endoscopic ultrasound (EUS) with synchronous fiducial marker placement and biopsy
* No evidence of distant metastases (M0)
* Medically fit to undergo surgical resection
* Life expectancy >6 months
* Adequate renal function to tolerate contrast dye for imaging
* ECOG Performance Status 0-2 Inclusion Criteria (Arm 1)
* Upfront resectable pancreatic cancer
* No evidence of nodal disease (N0)
* Appropriate to undergo a pancreaticoduodenectomy within 4-6 weeks of registration

Inclusion Criteria (Arm 2)

* Borderline resectable or upfront resectable pancreatic cancer
* Plan for surgical resection independent of the biochemical or radiographic response to SABR

Exclusion Criteria (Both Arms):

* Serious medical comorbidities or other contraindications to radiotherapy or surgery
* Gross disease involving duodenum or stomach
* Unable to have fiducials placed.
* Recurrent pancreatic cancer
* Prior abdominal radiation at any time
* Inability to attend full course of radiotherapy, surgery, or follow-up visits
* Contrast allergy
* Pregnant or lactating women

Exclusion Criteria (Arm 1):

* Receipt of any neoadjuvant system therapy, standard cytotoxic therapy or experimental

Exclusion Criteria (Arm 2):

* Elevated bilirubin or liver enzymes considered to be a contraindication to irinotecan chemotherapy, unless an intervention is planned to improve hepatic functioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity of Neoadjuvant SABR | 2 years
  Patients will be evaluated for toxicity during their follow-up exams according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Quality of Life (QOL) | 2 years
  QOL will be measured using the Functional Assessment of Cancer Therapy for Hepatobiliary and Pancreatic Subscale (FACT-Hep HCS)

SECONDARY OUTCOMES:
Change in tumor blood flow assessed by dynamic contrast enhanced CT imaging | <2 weeks after completion of chemotherapy (Arm 2 only)
  Dynamic Contrast enhanced CT imaging will be used to calculate tumor blood flow (ml^-1) within 2 weeks after completion of chemotherapy and calculate the change compared to baseline
Change in tumor blood flow assessed by dynamic contrast enhanced CT imaging | <6 hours after first fraction of radiation therapy (Arm 1 only)
  Dynamic Contrast enhanced CT imaging will be used to calculate tumor blood flow (ml^-1) within 6 hours after first fraction of radiation therapy and calculate the change compared to baseline
Change in tumor blood flow assessed by dynamic contrast enhanced CT imaging | <6 hours after first fraction of radiation therapy (Arm 2 only)
  Dynamic Contrast enhanced CT imaging will be used to calculate tumor blood flow (ml^-1) within 6 hours after first fraction of radiation therapy and calculate the change compared to that post-chemotherapy
Change in tumor blood flow assessed by dynamic contrast enhanced CT imaging | 2-4 weeks after radiation completed (Arm 1 only)
  Dynamic Contrast enhanced CT imaging will be used to calculate tumor blood flow (ml^-1) within 2-4 weeks after completion of radiation therapy and calculate the change compared to baseline
Change in tumor blood flow assessed by dynamic contrast enhanced CT imaging | 2-4 weeks after radiation completed (Arm 2 only)
  Dynamic Contrast enhanced CT imaging will be used to calculate tumor blood flow (ml^-1) 2-4 weeks after completion of radiation therapy and calculate the change compared to that post-chemotherapy
Predictive Value of Imaging Biomarkers of tumor metabolic uptake | 2 years
  Predictive value of 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG)-PET imaging biomarkers compared to pathologic outcome (complete response or non-complete response to treatment
Tumor recurrence | 2 years
  Time to local recurrence, regional recurrence, and distant recurrence of disease will be measured
Change in Cancer Antigen (CA) 19-9 expression | 2 years
  Change in CA19-9 detected in blood samples acquired before and after radiation therapy
Change in Carcinoembryonic antigen (CEA) expression | 2 years
  Change in CEA detected in blood samples acquired before and after radiation therapy
Detection of CD8+ T-cells | 2 years
  Peripheral blood samples will be evaluated using a plasma-based proteomics platform to detect T-cells after radiation therapy to examine peripheral markers of tumor immunity
Changes in markers of immune expression (CD3) | 2 years
  FFPE samples from pre-treatment biopsy tissue and post-treatment surgical resection samples to examine CD3 expression
Changes in markers of immune expression (CD8) | 2 years
  FFPE samples from pre-treatment biopsy tissue and post-treatment surgical resection samples to examine CD8 expression
Changes in markers of immune expression (PD-L1) | 2 years
  FFPE samples from pre-treatment biopsy tissue and post-treatment surgical resection samples to examine PD-L1 expression
Downstaging Rate (Arm 2) | 2-4 weeks post SABR
  Arm 2 patients will be re-evaluated for surgical resection. The ratio of the number of patients who proceed to surgery to the total number of patients that receive neoadjuvant FOLFIRINOX + SABR will be determined and subsequent therapy will be decided.
Negative Margin Resection Rate | Immediately post surgery
  Arm 1 patients (rPC) will be evaluated to ensure they remain fit for surgery. R0 vs. R1 resection will be determined and subsequent therapy will be decided. R0 vs. R1 resection will also be determined for Arm 2 (BRCP) patients that receive resection and subsequent therapy will be decided.
True Pathological Complete Response (PCR) | 2 years
  For both arms, those who exhibit a lack of viable tumor after surgical resection (e.g. a pathologic complete response [pCR]), which will be reported as the patients with a complete response, divided by the total number of patients undergoing resection, with a 95% confidence interval (CI).

IPD SHARING:
Plan to Share IPD: Undecided